CLINICAL TRIAL: NCT06663852
Title: Machine Learning-Based Decision Model for Optimal Adjuvant Therapy in Primary Gastric Neuroendocrine Carcinoma: a National Real-World Evidence Study
Brief Title: ML Decision Model for G-NEC Adjuvant Therapy
Acronym: G-NEC
Status: Completed | Type: Observational
Sponsor: Chang-Ming Huang, Prof. (Other)
Responsible Party: Sponsor-Investigator, Chang-Ming Huang, Prof., Prof., Fujian Medical University
Organization: Fujian Medical University (Other)
Other Study IDs: 2024GNEC
Record Dates: First submitted 2024-10-26; First posted 2024-10-29 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-10

CONDITIONS: Gastric Neuroendocrine Carcinoma (G-NEC); Postoperative Adjuvant Therapy for G-NEC; Survival Outcomes; Machine Learning
Keywords: Gastric Neuroendocrine Carcinoma (G-NEC); Adjuvant Chemotherapy; Machine Learning; Decision Support Model; Random Survival Forest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Gastric Neuroendocrine Carcinoma (G-NEC) Patients: This study focuses on patients diagnosed with gastric neuroendocrine carcinoma (G-NEC) who have undergone radical surgery. The cohort includes adult patients (≥18 years) treated at 38 tertiary hospitals in China between January 2006 and December 2020. Patients are divided into three groups based on their postoperative adjuvant treatment: no adjuvant chemotherapy, etoposide and platinum derivatives-based chemotherapy, and fluorouracil-based chemotherapy. The study aims to develop and validate a machine learning-based decision support model to optimize individualized adjuvant therapy strategies for G-NEC patients, with the primary outcome being disease-free survival (DFS).

SUMMARY:
Gastric neuroendocrine carcinoma (G-NEC) is a rare and aggressive tumor originating from neuroendocrine cells in the stomach lining. It is characterized by a high propensity for recurrence and a generally poor prognosis. Due to its rarity, there is limited data and no established consensus on the optimal postoperative adjuvant therapy, making treatment decisions challenging for healthcare providers.

This study is a retrospective analysis focusing on evaluating survival rates, identifying prognostic factors, and formulating treatment recommendations for patients with G-NEC. By analyzing real-world clinical data, we aim to better understand the factors that influence patient outcomes and to develop evidence-based strategies for improving survival. Our goal is to provide clinicians with valuable insights and tools to make more informed treatment decisions, ultimately enhancing the quality of care and outcomes for patients with this challenging disease.

ELIGIBILITY:
Inclusion Criteria:

* (1) patients who underwent radical surgery without any neoadjuvant therapy;
* (2) pathology confirmed NEC or mixed adenoneuroendocrine carcinoma (MANEC).

Exclusion Criteria:

* (1) history of other malignant neoplasms;
* (2) treatment with endoscopic submucosal dissection or endoscopic mucosal resection or thoracotomy;
* (3) incomplete clinical data (including pathological, adjuvant chemotherapy, and follow-up information);
* (4) receipt of alternative adjuvant treatment regimens;
* (5) death within 30 days postoperatively.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study includes adult patients diagnosed with gastric neuroendocrine carcinoma (G-NEC) or mixed adenoneuroendocrine carcinoma (MANEC) who underwent radical surgery at 38 tertiary hospitals in China between January 2006 and December 2020. The study population consists of patients who received either no adjuvant chemotherapy, etoposide and platinum derivatives-based chemotherapy, or fluorouracil-based chemotherapy following surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1505 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Disease-Free Survival (DFS) | From date of surgery up to 5 years
  Disease-free survival is defined as the time from the date of surgery to disease recurrence, death from any cause, or last follow-up, whichever occurs first. The machine learning model's performance in predicting DFS and recommending optimal adjuvant therapy will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided
Patient Privacy: As this study involves sensitive medical information, we must ensure that any data sharing plan complies with all relevant privacy laws and regulations.
  Ethical Considerations: We are consulting with our ethics committee to determine the most appropriate approach to data sharing that respects patient consent and maintains the integrity of the research.
  Data Standardization: Given the multi-center nature of this study, we are working on standardizing our data collection and storage processes across all 38 participating hospitals to ensure consistency and quality of any potentially shared data.
  Collaborative Potential: We recognize the value of data sharing in advancing gastric neuroendocrine carcinoma research and are exploring potential collaborations with other research groups.
  Resource Allocation: We are assessing the resources required to prepare the data for sharing, including de-identification processes and creation of data dictionaries.